CLINICAL TRIAL: NCT00263575
Title: A Multiple-Dose, Non-Randomized, Open-Label, Multicenter Study to Evaluate the Long-Term Safety and Effectiveness of EN3267 in the Treatment of Breakthrough Pain in Cancer Patients
Brief Title: Long-term Safety Study of Sublingual Fentanyl Tablets in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3267-007
Record Dates: First submitted 2005-12-07; First posted 2005-12-09 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Pain; Cancer
Keywords: EN3267; Breakthrough Pain; Safety Study; Fentanyl Tablets
MeSH Terms: conditions — Pain; Neoplasms; Breakthrough Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sublingual fentanyl tablet (Experimental)
  Interventions: Drug: EN3267

INTERVENTIONS:
Drug: EN3267 — EN3267 will be available in 100, 200, 300, 400, 600 (two 300 ug tablets), and 800 ug (two 400 ug tablets) doses
  Other Names: Fentanyl

SUMMARY:
The purpose of this study is to evaluate the long-term safety and effectiveness of EN3267 in treating breakthrough pain episodes in opioid cancer patients who are using stable doses of opioid medication.

DETAILED DESCRIPTION:
This was a Phase 3 non-randomized, open-label, multicentre study designed to evaluate the long-term safety of EN3267 in the treatment of BTcP in opioid-tolerant cancer patients. The study was conducted in 2 parts:

1. A Titration Period during which patients had up to 2 weeks to determine a single, effective dose of study medication (EN3267) for adequate treatment of BTcP, and
2. A maintenance Period of up to 12 months in which episodes of BTcP were treated with study medication.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 17 years of age or older.
* Stable cancer-related pain.
* Are receiving a stable, fixed-schedule oral opioid regimen equivalent to 60 to 1000 mg of oral morphine per day or transdermal fentanyl therapy equivalent to 50 to 300 µg/h, and are on a stable dose of opioid medication for relief of breakthrough pain.
* Experiencing 1-4 episodes of breakthrough pain per day.
* Meet the criteria defined in the Eastern Cooperative Oncology Group (ECOG) Performance Status for Grade 0, 1, or 2.

Exclusion Criteria:

* Have previously been exposed to EN3267.
* Are pregnant or lactating.
* Have uncontrolled or rapidly escalating pain.
* Have any clinically significant condition that would, in the investigator's opinion, preclude participation in the study or compromise data collection. These conditions may include cardiopulmonary disease, and/or neurologic/psychologic conditions.
* Are scheduled to take MAOIs (monoamine oxidase inhibitors) during the study.
* Are scheduled to receive anti-neoplastic therapy that, in the investigator's opinion, will influence assessment of breakthrough pain.
* Are scheduled to receive an investigational drug other than EN3267 during the course of the study.
* Have hypersensitivity, allergy or contraindication to fentanyl.
* Have significant prior history of substance abuse or alcohol abuse.
* Would have difficulty complying with the protocol, as assessed by the investigator.
* Are unable to read, write, or comprehend the English language in order to complete diaries.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Howell, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Carolinas Pain Institute, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Nalamachu S, Hassman D, Wallace MS, Dumble S, Derrick R, Howell J. Long-term effectiveness and tolerability of sublingual fentanyl orally disintegrating tablet for the treatment of breakthrough cancer pain. Curr Med Res Opin. 2011 Mar;27(3):519-30. doi: 10.1185/03007995.2010.545380. Epub 2011 Jan 6. PMID 21208151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was first patient screened in December 2005 to last patient screened in November 2008.
  Patients were recruited from Medical Institutions in the US.
Pre-assignment Details: Patients with stable cancer-related pain receiving stable, fixed-schedule oral opioid regimen. Patients were not permitted to have 2 consecutive days without at least 1 episode of BTcP. This regimen was for 14 days prior to screening and was expected to remain unchanged for the titration period. Patients with ulcerative mucositis were permitted.
Groups:
- Sublingual Fentanyl Tablet: EN3267 : EN3267 will be available in 100, 200, 300, 400, 600 (two 300 ug tablets), and 800 ug (two 400 ug tablets) doses
Period: Titration Period
Arm/Group | Sublingual Fentanyl Tablet
Started | 139
Completed | 96
Not Completed | 43
Not completed — Adverse Event | 14
Not completed — Withdrawal by Subject | 10
Not completed — Protocol Violation | 9
Not completed — Sponsor Decision | 2
Not completed — Other | 2
Not completed — Lack of Efficacy | 6
Period: Maintence Period
Arm/Group | Sublingual Fentanyl Tablet
Started | 96
Completed | 19
Not Completed | 77
Not completed — Adverse Event | 23
Not completed — Withdrawal by Subject | 8
Not completed — Protocol Violation | 4
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 6
Not completed — Lost to Follow-up | 1
Not completed — Sponsor Decision | 24
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Arm/Group | Sublingual Fentanyl Tablet
Number analyzed (Participants) | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 106
  >=65 years | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 63
Region of Enrollment [Number; unit: participants]
  United States | 139

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Long-term Safety and Effectiveness of EN3267
Time Frame: screening, 2 week titration period and 12 monthly study visits
Measure: Number; unit: participants
Groups:
- Titration: EN3267: EN3267 will be available in 100, 200, 300, 400, 600 (two 300 ug tablets), and 800 ug (two 400 ug tablets) doses
- Maintenance: All patients enrolled who continued into the maintenance period
- Overall: Combination of titration and maintenance period
Arm/Group | Titration | Maintenance | Overall
Number analyzed (Participants) | 139 | 96 | 139
participants
  Patients with at least 1 AE | 64 | 87 | 116
  Patients with at least 1 AE causing discontinue | 14 | 23 | 37
  Patients with at least 1 SAE | 7 | 40 | 46
  Patients with an AE resulting in death | 4 | 15 | 19

ADVERSE EVENTS:
Arm/Group | Sublingual Fentanyl Tablet
Serious Adverse Events (participants affected / at risk) | 46/139
Other Adverse Events (participants affected / at risk) | 116/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sublingual Fentanyl Tablet (N=139)
death (General disorders) | 19
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Esophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Central line infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Candida sepsis (Infections and infestations) | 1
Intestinal fistula infection (Infections and infestations) | 1
Pneumonia herpes viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Anemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 2
Coagulopathy (Blood and lymphatic system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructed airway disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 1
Pain (General disorders) | 3
Asthenia (General disorders) | 1
Infusion site reaction (General disorders) | 1
Convulsion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Azotemia (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Obstructive uropathy (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Immunosuppression (Immune system disorders) | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sublingual Fentanyl Tablet (N=139)
Nausea (Gastrointestinal disorders) | 32
Vomiting (Gastrointestinal disorders) | 18
Constipation (Gastrointestinal disorders) | 12
Diarrhea (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 21
Edema peripheral (General disorders) | 15
Asthenia (General disorders) | 12
Somnolence (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 9
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 13
Weight decreased (Investigations) | 8
Rash (Skin and subcutaneous tissue disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 16
Anorexia (Metabolism and nutrition disorders) | 11
Hypokalemia (Metabolism and nutrition disorders) | 7
Anemia (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Insomnia (Psychiatric disorders) | 13
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 8
Hypotension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication statement in clinical trial agreement